CLINICAL TRIAL: NCT00282243
Title: A Phase 2, Open-Label, Multi-Center Study to Assess the Pharmacokinetics, Long-term Safety and Tolerability of Tacrolimus in Stable Liver Transplant Patients Converted From a Prograf® Based Immunosuppression Regimen to a Modified Release (MR) Tacrolimus Based Immunosuppression Regimen
Brief Title: A Study to Assess the Pharmacokinetics of a Modified-release Tacrolimus Based Immunosuppression Regimen in Stable Liver Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02-0-152
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-08

CONDITIONS: Liver Transplantation
Keywords: Pharmacokinetics; Therapy; Immunosuppression; Drugs, Investigational; Adult
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus MR (Experimental): After enrollment in the pharmacokinetic period, patients were maintained on their usual dose of tacrolimus twice daily on Day 1 through Day 14 and on Day 15 were converted to tacrolimus modified release (MR) once-daily in the morning for 14 days, converted back to tacrolimus twice daily for 14 days and then converted back to tacrolimus MR formulation once-daily in the morning for 14 days, all based on a 1:1 mg for mg total daily dose conversion. The extended treatment period began on day 57 and consisted of a single dose of tacrolimus extended-release formulation once every morning through the end of the study.
  Dose adjustments were allowed in order to maintain the target tacrolimus trough level within the range of 5 to 20 ng/mL and for clinical reasons.
  Interventions: Drug: tacrolimus modified release (MR); Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus modified release (MR) — Oral
  Other Names: Advagraf,; FK506E,; MR4,; FKMR,; Astagraf XL
Drug: tacrolimus — Oral
  Other Names: Prograf,; FK506

SUMMARY:
A study to assess the pharmacokinetics, safety and effectiveness of tacrolimus in stable liver transplant patients converted from a tacrolimus (Prograf®) based immunosuppression regimen to a modified release tacrolimus based immunosuppression regimen.

DETAILED DESCRIPTION:
A one arm study to assess the pharmacokinetics, safety and effectiveness of tacrolimus in stable liver transplant patients converted from a tacrolimus (Prograf®) based immunosuppression regimen to a modified release tacrolimus based immunosuppression regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently receiving Prograf ® based immunosuppressive therapy for liver transplantation.
* Patient has stable whole blood trough level concentrations of Prograf® and is clinically stable

Exclusion Criteria:

* Patient has previously received an organ transplant other than a liver
* Patient is currently receiving sirolimus immunosuppression therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (10):
- United States (10):
  - Palo Alto, California
  - Denver, Colorado
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - New York, New York
  - Cincinnati, Ohio
  - Dallas, Texas
  - Madison, Wisconsin

REFERENCES:
- [Background] Florman S, Alloway R, Kalayoglu M, Punch J, Bak T, Melancon J, Klintmalm G, Busque S, Charlton M, Lake J, Dhadda S, Wisemandle K, Wirth M, Fitzsimmons W, Holman J, First MR. Once-daily tacrolimus extended release formulation: experience at 2 years postconversion from a Prograf-based regimen in stable liver transplant recipients. Transplantation. 2007 Jun 27;83(12):1639-42. doi: 10.1097/01.tp.0000265445.09987.f1. PMID 17589349
- [Background] Florman S, Alloway R, Kalayoglu M, Lake K, Bak T, Klein A, Klintmalm G, Busque S, Brandenhagen D, Lake J, Wisemandle K, Fitzsimmons W, First MR. Conversion of stable liver transplant recipients from a twice-daily Prograf-based regimen to a once-daily modified release tacrolimus-based regimen. Transplant Proc. 2005 Mar;37(2):1211-3. doi: 10.1016/j.transproceed.2004.11.086. PMID 15848672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stable liver transplant recipients aged 18 to 65 years who were on a stable dose of tacrolimus based immunosuppressive regimen.
Pre-assignment Details: Pharmacokinetic (PK) treatment period was 56 days. Participants who completed the PK period were eligible to continue receiving tacrolimus MR in the extended treatment period, from Day 57 up to 60 months.
Period: Pharmacokinetic Treatment Period
Arm/Group | Tacrolimus MR
Started | 70
Received Tacrolimus | 70
Received Tacrolimus MR | 69
Completed | 65
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Period: Extension Treatment Period
Arm/Group | Tacrolimus MR
Started | 65
Completed | 43
Not Completed | 22
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 4
Not completed — Non-compliance | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic evaluable set, defined as all patients with four complete pharmacokinetic profiles (two tacrolimus and two tacrolimus MR).
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 50.3 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  White | 57
  Black | 4
  Pacific Islander | 1
Reason for End Stage Liver Disease [Number; unit: participants]
  Hepatitis C | 15
  Alcoholic Liver Disease | 11
  Autoimmune Disease | 4
  Primary Biliary Cirrhosis | 7
  Primary Sclerosing Cholangitis | 6
  Alpha-1 Anti-Trypsin Deficiency | 3
  Hepatitis B | 2
  Non-Alcoholic Steatohepatitis | 2
  Cryptogenic Cirrhosis | 2
  Unknown | 1
  Other | 9
Type of Current Transplant [Number; unit: participants]
  Whole Cadaver | 56
  Living related Donor | 3
  Split Cadaver | 3
Re-transplant [Number; unit: participants]
  No | 56
  Yes | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) for Tacrolimus
Description: The area under the concentration-time curve was calculated from whole blood tacrolimus concentrations for both the tacrolimus and tacrolimus MR treatment periods at steady state using the linear trapezoidal rule. The AUC0-24 for tacrolimus was calculated as the sum of the AUC0-12 for the morning (0-12 hour) and afternoon (12-24 hour) doses.
Time Frame: Days 14 and 42 (tacrolimus) and Days 28 and 56 (tacrolimus MR), pre-dose 0.5, 1, 2, 3, 4, 6, 8, 12 (pre-dose for tacrolimus only), 12.5, 13, 14, 15, 16, 18, 20, and 24 hours post-dose.
Population: Pharmacokinetic evaluable set defined as all patients with four complete pharmacokinetic profiles (two tacrolimus and 2 tacrolimus MR).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 62
ng*hr/mL
  Day 14: Tacrolimus | 215.6 (77.8)
  Day 28: Tacrolimus MR | 184.0 (62.7)
  Day 42: Tacrolimus | 202.4 (53.3)
  Day 56: Tacrolimus MR | 187.9 (58.1)
Statistical Analysis 1: Comparison: Tacrolimus MR; The method of analysis of variance with repeated measures was used for the comparisons of AUC0-24. Exposure at steady state was used for tacrolimus (steady state was defined as days 14 and 42) and for tacrolimus MR (steady state was defined as days 28 and 56). The natural log (ln) was used to transform AUC0-24 prior to analysis and the results were transformed back to the original scale for the presentation of results; Test type: Non-Inferiority or Equivalence — If the 90% CI for the ratio of the natural log-transformed pharmacokinetic parameters fell within an 80% to 125% range, then the exposure between the two formulations was considered to be equivalent; Ratio of means = 88.79, 90% CI 2-sided [85.42 to 92.29] — Tacrolimus/tacrolimus MR ratio of natural log transformed means expressed as a percent

2. Secondary Outcome: Maximum Observed Concentration of Tacrolimus (Cmax)
Description: The maximum concentration was calculated from whole blood tacrolimus concentrations for both the tacrolimus and tacrolimus MR treatment periods at steady state, without interpolation.
Time Frame: Days 14 and 42 (tacrolimus) and Days 28 and 56 (tacrolimus MR), pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 (pre-dose for tacrolimus only), 12.5, 13, 14, 15, 16, 18, 20, and 24 hours post-dose.
Population: Pharmacokinetic evaluable set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 62
ng/mL
  Day 14: Tacrolimus | 17.9 (9.9)
  Day 28: Tacrolimus MR | 13.3 (5.6)
  Day 42: Tacrolimus | 16.0 (6.9)
  Day 56: Tacrolimus MR | 14.1 (6.0)

3. Primary Outcome: Minimum Observed Concentration of Tacrolimus (Cmin)
Description: The trough (minimum) concentration of tacrolimus determined from the tacrolimus whole blood concentration value at the 12 hour post-dose concentration based on the evening dose (i.e., the 8 am concentration) for tacrolimus and the 24-hour time point post-dose for tacrolimus MR, prior to receiving the next dose.
Time Frame: Days 14 and 42 at 12 hours post-dose (tacrolimus) and Days 28 and 56 at 24 hours post-dose (for tacrolimus MR).
Population: Pharmacokinetic evaluable set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 62
ng/mL
  Day 14: Tacrolimus | 7.1 (2.5)
  Day 28: Tacrolimus MR | 5.5 (1.8)
  Day 42: Tacrolimus | 6.8 (1.8)
  Day 56: Tacrolimus MR | 5.8 (1.8)
Statistical Analysis 1: Comparison: Tacrolimus MR; The method of analysis of variance with repeated measures was used for the comparisons of Cmin. Exposure at steady state was used for tacrolimus (steady state was defined as days 14 and 42) and for tacrolimus MR (steady state was defined as days 28 and 56). The natural log (ln) was used to transform Cmin prior to analysis and the results were transformed back to the original scale for the presentation of results; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of means = 81.40, 90% CI 2-sided [77.88 to 85.08] — Tacrolimus/tacrolimus MR ratio of natural log transformed means expressed as a percent

4. Primary Outcome: Patient Survival
Description: Patient survival was defined as any participant known to be alive at the time of analysis.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set, defined as all patients who took at least one dose of tacrolimus MR during the extended treatment period of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 65
percentage of participants | 92.31 [85.83 to 98.79]

5. Primary Outcome: Graft Survival
Description: Graft survival was defined as any participant who did not meet the definition of graft loss, where graft loss was defined as graft failure (re-transplant) or participant death.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 65
percentage of participants | 90.77 [83.73 to 97.81]

6. Secondary Outcome: Time to Maximum Observed Concentration of Tacrolimus (Tmax)
Description: Time to the first occurrence to reach the maximum concentration of tacrolimus was calculated from whole blood tacrolimus concentrations for both the tacrolimus and tacrolimus MR treatment periods at steady state, without interpolation.
Time Frame: as for outcome 2
Population: Pharmacokinetic evaluable set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 62
hours
  Day 14: Tacrolimus | 2.8 (4.2)
  Day 28: Tacrolimus MR | 3.0 (3.1)
  Day 42: Tacrolimus | 3.0 (4.4)
  Day 56: Tacrolimus MR | 2.7 (2.1)

7. Secondary Outcome: Percentage of Participants With Biopsy-confirmed Acute Rejection
Description: Biopsy-confirmed acute rejection (BCAR) is defined as an episode of acute liver allograft rejection that was confirmed by biopsy results and was Banff grade ≥ I. Biopsies were graded by the pathologist at the clinical site according to the 1997 Banff criteria for grading of acute liver allograft rejection: Indeterminate: Portal inflammatory infiltrate that fails to meet the criteria for diagnosis of acute rejection; Grade I (Mild): Rejection infiltrate in a minority of the triads that is generally mild and confined within the portal spaces; Grade II (Moderate): Rejection infiltrate, expanding to most or all of the triads; Grade III (Severe): Rejection infiltrate, expanding to most or all of the triads, with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte necrosis.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 65
percentage of participants | 9.23 [2.19 to 16.27]

8. Secondary Outcome: Time to Event for Patient Non-survival
Description: For participants who died on study, the median number of days from first dose of study drug to death due to any cause.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set who died on study.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 5
days | 1561.00 [720.0 to 1881.0]

9. Secondary Outcome: Time to Event for Graft Non-survival
Description: For participants with graft loss, the median number of days from the first dose of study drug to graft loss. Graft loss was defined as graft failure (re-transplant) or participant death.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with graft loss.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 6
days | 1529.50 [720.0 to 1881.0]

10. Secondary Outcome: Time to First Biopsy-confirmed Acute Rejection
Description: For participants with a biopsy-confirmed acute rejection (BCAR), the median number of days from the first dose of study drug to the date of biopsy confirmation. BCAR is defined as an episode of acute liver allograft rejection that was confirmed by biopsy results and was Banff grade ≥ I. Biopsies were graded by the clinical site pathologist according to the 1997 Banff criteria for grading acute liver allograft rejection: Indeterminate: Portal inflammatory infiltrate that fails to meet the criteria for diagnosis of acute rejection; Grade I: Rejection infiltrate in a minority of the triads that is generally mild and confined within the portal spaces; Grade II: Rejection infiltrate, expanding to most or all of the triads; Grade III: Rejection infiltrate, expanding to most or all of the triads, with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte necrosis.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with a biopsy-confirmed acute rejection.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 6
days | 802.50 [153.0 to 1871.0]

11. Secondary Outcome: Grade of Biopsy-confirmed Acute Rejection Episodes
Description: Biopsy-confirmed acute rejection (BCAR) is defined as an episode of acute liver allograft rejection that was confirmed by biopsy results and was Banff grade ≥ I. Biopsies were graded by the clinical site pathologist according to the 1997 Banff criteria for grading of acute liver allograft rejection: Indeterminate: Portal inflammatory infiltrate that fails to meet the criteria for diagnosis of acute rejection; Grade I (Mild): Rejection infiltrate in a minority of the triads that is generally mild and confined within the portal spaces; Grade II (Moderate): Rejection infiltrate, expanding to most or all of the triads; Grade III (Severe): Rejection infiltrate, expanding to most or all of the triads, with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte necrosis. For participants with more than one biopsy-confirmed acute rejection episode, the worst case grade is reported.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with a biopsy-confirmed acute rejection.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 6
participants
  Grade I | 4
  Grade II | 2
  Grade III | 0

12. Secondary Outcome: Number of Participants Receiving Anti-lymphocyte Antibody Therapy for Acute Rejection
Description: Steroid-resistant rejection episodes were treated with anti-lymphocyte antibodies. If a participant had a histologically proven Banff Grade II or III rejection, they could be initiated on anti-lymphocyte antibody treatment per institutional practice.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 65
participants | 1

13. Secondary Outcome: Number of Participants With Multiple Rejection Episodes
Description: This analysis includes rejection episodes that were either confirmed by biopsy by the clinical site pathologist or were clinically treated.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 65
participants | 2

14. Secondary Outcome: Number of Participants With Clinically Treated Acute Rejection Episodes
Description: A clinically treated acute rejection episode was any biopsy-confirmed or suspected rejection episode that was treated with immunosuppressive therapy.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 65
participants | 5

15. Secondary Outcome: Number of Participants With Chronic Rejection
Description: Due to the low number of participants with biopsy-confirmed acute rejection episodes, chronic rejection was not analyzed.
Time Frame: From enrollment until the end of study (up to 60 months).
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure was defined as discontinuation of study drug for any reason. Due to discontinuation of the study by the sponsor, treatment failure was not analyzed.
Time Frame: From enrollment until the end of study (up to 60 months).
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 0

17. Secondary Outcome: Primary Reason for Graft Loss
Description: The primary reason for graft loss was recorded by the Investigator. Graft loss was defined as graft failure (re-transplant) or participant death.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with graft loss.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 6
participants
  Recurrent disease | 1
  Death | 5

18. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: Hepatic function was assessed by measuring alanine aminotransferase levels over the course of the study.
Time Frame: Baseline (the last day of tacrolimus on Day 14 prior to the first conversion to tacrolimus MR), Day 56 (end of the pharmacokinetic phase) and end of treatment (EOT; the last observed value during treatment, maximum time on study was 60 months).
Population: Modified safety analysis set defined as all patients who took at least 1 dose of tacrolimus and at least one dose of tacrolimus MR during the pharmacokinetic portion of the study. "N" indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 69
U/L
  Baseline [N= 69] | 38.5 (22.38)
  Change from Baseline at Day 56 [N=67] | 14.4 (79.16)
  Change from Baseline at EOT [N=68] | 13.3 (60.60)

19. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST)
Description: Hepatic function was assessed by measuring aspartate aminotransferase levels over the course of the study.
Time Frame: as for outcome 18
Population: Modified safety analysis set. "N" indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 69
U/L
  Baseline [N= 69] | 33.4 (17.94)
  Change from Baseline at Day 56 [N=67] | 3.6 (23.32)
  Change from Baseline at EOT [N=68] | 10.6 (55.05)

20. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Hepatic function was assessed by measuring total bilirubin over the course of the study.
Time Frame: as for outcome 18
Population: Modified safety analysis set. "N" indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 69
mg/dL
  Baseline [N= 69] | 0.74 (0.604)
  Change from Baseline at Day 56 [N=67] | 0.03 (0.657)
  Change from Baseline at EOT [N=68] | 1.04 (5.948)

21. Secondary Outcome: Safety as Assessed by Adverse Events, Laboratory Parameters and Vital Signs
Description: An adverse event is defined as any reaction, side effect or other untoward medical occurrence, regardless of the relationship to study drug which occurred during the conduct of a clinical study. Clinically significant adverse changes in clinical status, routine laboratory studies or physical examinations were considered adverse events.
  A serious adverse event was any adverse event occurring at any dose that resulted in any of the following outcomes:
  * Death
  * Life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability or incapacity
  * Congenital abnormality or birth defect
  * Important medical event.
Time Frame: From the first dose of tacrolimus MR formulation through the last dose day plus 10 days (approximately 60 months).
Population: Modified safety analysis set.
Measure: Number; unit: participants
Arm/Group | Tacrolimus MR
Number analyzed (Participants) | 69
participants
  Any adverse event | 63
  Serious adverse event | 37
  Adverse event leading to discontinuation | 18
  Adverse event leading to dose changes | 37
  Death | 5

ADVERSE EVENTS:
Time Frame: From the first dose of tacrolimus MR formulation through the last dose day plus 10 days (approximately 60 months).
Description: Adverse events are reported for the modified safety analysis set defined as all patients who took at least 1 dose of tacrolimus and one dose of tacrolimus MR during the pharmacokinetic period of the study.
Arm/Group | Tacrolimus MR
Serious Adverse Events (participants affected / at risk) | 37/69
Other Adverse Events (participants affected / at risk) | 51/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus MR (N=69)
Pneumonia (Infections and infestations) | 5
Influenza (Infections and infestations) | 2
Bronchiectasis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Enterobacter sepsis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Haemobilia (Hepatobiliary disorders) | 1
Hepatitis granulomatous (Hepatobiliary disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 4
Postoperative haematoma (Injury, poisoning and procedural complications) | 2
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Postoperative heterotopic calcification (Injury, poisoning and procedural complications) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Unspecified malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial fibrillation (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypolycaemia (Metabolism and nutrition disorders) | 1
Renal failure acute (Renal and urinary disorders) | 6
Acute prerenal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Renal insufficiency (Renal and urinary disorders) | 1
Pyrexia (General disorders) | 4
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Hernia (General disorders) | 1
Rigors (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Graft loss (Immune system disorders) | 1
Liver transplant rejection (Immune system disorders) | 1
Transplant rejection (Immune system disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Blood creatinine increased (Investigations) | 1
International normalized ratio increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Aphasia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Disorientation (Psychiatric disorders) | 1
Drug dependence (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Spinal laminectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus MR (N=69)
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 6
Influenza (Infections and infestations) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Renal impairment (Renal and urinary disorders) | 9
Renal insufficiency (Renal and urinary disorders) | 7
Blood creatinine increased (Investigations) | 6
Liver function test abnormal (Investigations) | 6
Hepatic enzyme increased (Investigations) | 4
Headache (Nervous system disorders) | 13
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Hypertension (Vascular disorders) | 8
Fatigue (General disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or until 18 months have elapsed following study completion. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document.